CLINICAL TRIAL: NCT06313268
Title: Post-marketing Safety of Effivia®, a Bevacizumab Biosimilar: Phase IV, Observational, Multicenter Clinical Study in Mexican Population
Brief Title: Safety of Effivia®, a Bevacizumab Biosimilar
Status: Completed | Type: Observational
Sponsor: Laboratorios Liomont (Industry)
Collaborators: Servicios Especializados en Ensayos Clínicos, S.C. (Unknown)
Responsible Party: Sponsor
Other Study IDs: LT-02-20
Record Dates: First submitted 2024-02-21; First posted 2024-03-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Cancer; Metastatic Cervical Cancer; Non Squamous Non Small Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Test group: Bevacizumab (Effivia®)
  Interventions: Drug: Bevacizumab Biosimilar MB02

INTERVENTIONS:
Drug: Bevacizumab Biosimilar MB02 — 5 mg/kg to 15 mg/kg in combination with chemotherapy.
  Other Names: Effivia®

SUMMARY:
This is a post-marketing observational study aimed to evaluated the safety profile of Effivia®, a biosimilar of bevacizumab, in mexican patients with different types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 18 years and older.
* Patients with metastatic colorectal cancer,unresectable, locally advanced, recurrent or metastatic non-squamous non-small cell lung cancer, metastatic renal cell carcinoma, persistent, recurrent, or metastatic cervical cancer, or epithelial ovarian, fallopian tube, or primary peritoneal cancer naive to bevacizumab therapy (Effivia®).
* Provide written informed consent.

Exclusion Criteria:

* History of recent surgery or wound healing complications.
* History of gastrointestinal perforations or fistula.
* History of renal injury and proteinuria.
* Recent surgical intervention.
* Pregnant or nursing women.
* History of bevacizumab, monoclonal antibodies, or CHO cells-derived products hypersensitivity.
* Other safety concerns or bevacizumab contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Naive to bevacizumab, adult patients with metastatic colorectal cancer, metastatic cervical cancer, non-squamous non-small cell lung cancer, and other cancer types where Bevacizumab therapy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Adverse events | From date of patient inclusion to the end of Cycle 1 (each cycle is up to six months)
  Frequency and characteristics of adverse events (serious and non serious)

CONTACTS AND LOCATIONS:
Locations (5):
- Mexico (5):
  - UMAE Hospital de Especialidades No. 1, León, Guanajuato
  - Hospital de Gineco-Obstetricia No. 3, Azcapotzalco, Mexico City
  - Hospital de Oncología, UMAE Centro Médico Nacional Siglo XXI, Cuauhtémoc, Mexico City
  - Instituto Nacional de Cancerología, Tlalpan, Mexico City
  - Hospital de Oncología IMSS Puebla, Puebla City

IPD SHARING:
Plan to Share IPD: No